CLINICAL TRIAL: NCT03454828
Title: Mechanisms of Obesity and Its Metabolic Complications in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000022239; 1R01DK114504-01A1 (NIH)
Record Dates: First submitted 2018-02-19; First posted 2018-03-06 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- obese carbohydrate diet (Experimental): Obese adolescents with a body mass index (BMI) >95th percentile.
  Interventions: Dietary Supplement: obese carbohydrate diet
- lean carbohydrate diet (Active Comparator): Lean adolescents with a body mass index (BMI) <85th percentile.
  Interventions: Dietary Supplement: lean carbohydrate diet

INTERVENTIONS:
Dietary Supplement: obese carbohydrate diet — The experimental diet will consist of 30% carbohydrates (CHO), 35% protein, and 35% fat. Since the experimental diet is lower in CHO, the fiber and sugar content will be calculated based on total CHO in the same percentage as the control (0.25 g fiber per each kcal of CHO and 18.2% sugar for total CHO).
  Arms: obese carbohydrate diet
Dietary Supplement: lean carbohydrate diet — The control diet composition will follow the American Dietary Guidelines of 55% carbohydrates (CHO), 15% protein, and 30% fat. CHO content will be primarily complex CHO of high quality (14 g fiber/1,000 kcals and <10% of total kcals in the form of sugar).
  Arms: lean carbohydrate diet

SUMMARY:
The overarching goal of this project is to determine whether the effect of gut microbiota on human metabolism might be mediated by short chain fatty acids (SCFA) and whether the SCFA might modulate lipid metabolism.

DETAILED DESCRIPTION:
This would be the first study determining the effect of SCFA synthesis on hepatic de novo lipogenesis and to assess whether and how isocaloric dietary changes (namely low carbohydrates) might modify the composition of the gut microbiota and reduce the synthesis of SCFA during adolescence, a sensitive period for the development of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Good general health,
* Taking no medication on a chronic basis
* Age 15 to 21 years,
* In puberty (girls and boys: Tanner stage III - V)
* BMI >25th and <85th for lean cohort; BMI >95th for obese cohort
* Girls who begin menstruating must have a negative pregnancy test during the study.

Exclusion criteria:

* Baseline creatinine >1.0 mg
* Food allergies
* Pregnancy
* Presence of endocrinopathies (e.g. Cushing syndrome)
* Significant chronic illness.

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2018-08-18 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Santoro, Phd,MD, Principal Investigator — Yale University
Locations (1):
- Hospital Research Unit, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Galuppo B, Umano GR, Li Z, Van Name M, Samuels SL, Kien CL, Cline GW, Wagner DA, Barbieri E, Trico D, Santoro N. Comparison of Metabolic Response to Colonic Fermentation in Lean Youth vs Youth With Obesity. JAMA Netw Open. 2023 May 1;6(5):e2312530. doi: 10.1001/jamanetworkopen.2023.12530. PMID 37159195
- [Derived] Galuppo B, Cline G, Van Name M, Shabanova V, Wagner D, Kien CL, Santoro N. Colonic Fermentation and Acetate Production in Youth with and without Obesity. J Nutr. 2021 Nov 2;151(11):3292-3298. doi: 10.1093/jn/nxab277. PMID 34494088
- [Derived] Monga Kravetz A, Testerman T, Galuppo B, Graf J, Pierpont B, Siebel S, Feinn R, Santoro N. Effect of Gut Microbiota and PNPLA3 rs738409 Variant on Nonalcoholic Fatty Liver Disease (NAFLD) in Obese Youth. J Clin Endocrinol Metab. 2020 Oct 1;105(10):e3575-85. doi: 10.1210/clinem/dgaa382. PMID 32561908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children and adolescents between 15 and 25 years of age.
Groups:
- Youth With Obesity: Obese adolescents with a body mass index (BMI) >95th percentile.
- Lean Youth: Lean adolescents with a body mass index (BMI) <85th percentile.
Period: Overall Study
Arm/Group | Youth With Obesity | Lean Youth
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The overall number of participants included in the baseline analysis population is less than the number of participants assigned to study arms because some participants did not complete baseline assessments or had missing baseline data
Groups:
- Total: Total of all reporting groups
Arm/Group | Youth With Obesity | Lean Youth | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 16 | 28
  Between 18 and 65 years | 7 | 3 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 14 | 18 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 0 | 8
  White | 6 | 17 | 23
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Rate of appearance of acetate [Mean (Standard Deviation); unit: μmol · kg-1 · min-1] | 7.40 (4.44) | 7.69 (7.541) | 7.55 (6.097)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Appearance of Acetate
Description: Starting at 08:00, we began a 10-h, primed, continuous, peripheral venous infusion of 99% sodium [d3]-acetate with a priming dose of 200 μg · kg-1 · min-1 for 4 min and a continuous infusion rate of 59.5 μg · kg-1 · min-1 for 10 h. After 180 min from the start of the infusion, subjects received 20 g of lactulose per os, dissolved in 30 mL of water.
Time Frame: Pre lactulose (average values at 2, 2.5, 3 hours) and Post lactulose (average of values at 7, 8, 9 and 10 hours)
Measure: Mean (Standard Error); unit: umol/kg/min
Arm/Group | Youth With Obesity | Lean Youth
Number analyzed (Participants) | 19 | 19
umol/kg/min
  Pre-lactulose | 7.40 (1.73) | 7.69 (1.02)
  Post-lactulose | 9.29 (1.44) | 14.7 (2.33)

2. Primary Outcome: Percent of Hepatic de Novo Lipogenesis.
Description: The percent of hepatic de novo lipogenesis (DNL) refers to the proportion of fatty acids in the liver that are derived from a de novo synthesis pathway, rather than from dietary sources.
Time Frame: Pre lactulose (average values at 2, 2.5, 3 hours) and Post lactulose (average of values at 7, 8, 9 and 10 hours)
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Youth With Obesity | Lean Youth
Number analyzed (Participants) | 6 | 5
Percentage
  Pre Lactulose | 1.96 (0.159) | 2.53 (0.364)
  Post Lactulose | 1.97 (0.192) | 3.38 (0.62)

3. Primary Outcome: Change in the Rate of Appearance of Acetate
Description: The changes in rate of appearance of acetate (RaAcetate) are measured averaging the basal RaAcetate 9 timepoints (2 and 3 hours) and the post-lactulose RaAcetate (timepoints 7, 8, 9 and 10 hours).
Time Frame: Pre lactulose (average values at 2, 2.5, 3 hours) and Post lactulose (average of values at 7, 8, 9 and 10 hours)
Measure: Mean (Standard Deviation); unit: micromol/Kg/minute
Groups:
- Low Carbohydrate Diet: Obese adolescents with a body mass index (BMI) >95th percentile.
  The experimental diet consisted of 30% carbohydrates (CHO), 35% protein, and 35% fat.
- Normal Carbohydrate Diet: Lean adolescents with a body mass index (BMI) <85th percentile.
  The normal diet composition followed the American Dietary Guidelines of 55% carbohydrates (CHO), 15% protein, and 30% fat. CHO content will be primarily complex CHO of high quality (14 g fiber/1,000 kcals and <10% of total kcals in the form of sugar).
Arm/Group | Low Carbohydrate Diet | Normal Carbohydrate Diet
Number analyzed (Participants) | 4 | 4
micromol/Kg/minute
  Pre Diet | -2.34 (6.57) | 1.63 (1.75)
  Post Diet | -1.59 (7.55) | -0.96 (6.76)
Statistical Analysis 1: Comparison: Low Carbohydrate Diet vs Normal Carbohydrate Diet; Test type: Superiority; p = 0.399, t-test, 2 sided; Mean Difference (Final Values) = 0.118

ADVERSE EVENTS:
Time Frame: 10 HOURS
Groups:
- Youth With Obesity or Overweight: Youth with a BMI percentile above 85th
- Youth Without Obesity: Youth with a BMI percentile below 75th
Arm/Group | Youth With Obesity or Overweight | Youth Without Obesity
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

LIMITATIONS AND CAVEATS:
The study included a relatively small cohort of participants, which may limit the statistical power and generalizability of the findings. Differences in gut microbiota composition were not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT03454828/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT03454828/ICF_001.pdf